CLINICAL TRIAL: NCT02489227
Title: A Double-Blind, Randomized, Parallel-Group, Active-Control Study to Compare the Efficacy and Safety of CHS-1420 Versus Humira in Subjects With Chronic Plaque Psoriasis
Brief Title: Comparison of CHS-1420 Versus Humira in Subjects With Chronic Plaque Psoriasis
Acronym: PsOsim
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Coherus Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHS-1420-02
Record Dates: First submitted 2015-07-01; First posted 2015-07-02 (Estimated); Results first posted 2019-10-18 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Plaque Psoriasis
Keywords: PsO
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Humira (adalimumab) (Active Comparator): Adalimumab (Humira) 40mg 2 doses at week 0/Day 0, then 1 dose every 2 weeks starting at Week 1 until Week 15. At Week 16 subjects initially randomized to adalimumab will be assigned (1:1) to CHS-1420 or continue adalimumab treatment, 1 dose every 2 weeks for weeks 17-23. The assignments for treatment sequences (Treatment Period 1 and Treatment Period 2) were made randomly at the beginning of Treatment Period 1. At week 24 subjects will switch to CHS-1420 open label until study end.
  Interventions: Drug: CHS-1420; Drug: Adalimumab
- CHS-1420 (Experimental): CHS-1420 40mg 2 doses at Week 0/Day 0 then 1 dose every 2 weeks starting at Week 1 for 23 weeks. At Week 24 subjects will continue on to CHS-1420 open label until study end.
  Interventions: Drug: CHS-1420

INTERVENTIONS:
Drug: CHS-1420
Drug: Adalimumab
  Other Names: Humira
  Arms: Humira (adalimumab)

SUMMARY:
This is a 3-period study comparing CHS-1420 to Humira in patients with chronic plaque psoriasis.

DETAILED DESCRIPTION:
This is a 55-week, randomized, double-blind, active-control, parallel group, multicenter, global study in subjects with active, moderate to severe, chronic PsO.

The study will consist of 24 weeks of administration of blinded study drug, divided into Treatment Period 1 and Treatment Period 2, then 23 weeks of administration of open-label CHS-1420 and a Follow-up visit 8 weeks after the last dose. Subjects who meet inclusion/exclusion criteria will be stratified by body mass index (BMI), and age and randomized 1:1 to receive CHS-1420 or Humira in Treatment Period 1. Subjects assigned to CHS-1420 will continue to receive CHS-1420 in Period 2. Subjects assigned to Humira in Period 1 will be randomly assigned (1:1) to either continue with Humira in Treatment Period 2 or to switch to CHS-1420 in Treatment Period 2. All subjects will receive open label CHS-1420 in Treatment Period 3.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults
* PsO diagnosis for 6 months
* Active disease: PASI greater than or equal to 12, Physician's Static Global Assessment (PSGA) score greater than or equal to 3 (based on a scale of 0-5),
* Body Surface Area (BSA) involved with PsO greater than or equal to 10%

Exclusion Criteria:

* Forms of psoriasis other than PsO
* Drug induced psoriasis
* Positive QuantiFERON-tuberculosis (TB) Gold Test
* Presence of significant comorbid conditions
* Chemistry and hematology values outside protocol specified range
* Major systemic infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05-06 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara P Finck, M.D., Study Director — Coherus Oncology, Inc.
Locations (98):
- United States (28):
  - Sadra Sasha Jazayeri, MD, Phoenix, Arizona
  - Encino Research Center, Encino, California
  - Center for Dermatology and Laser Surgery, Sacramento, California
  - Kenneth M Stein, MD, Santa Rosa, California
  - HealthCare Partners Medical Group Clinical Research Center, Torrance, California
  - Horizons Clinical Research Center, LLC., Denver, Colorado
  - New England Research Associates LLC, Trumbull, Connecticut
  - Francisco A Kerdel, MD, Coral Gables, Florida
  - Linda Tripodis Murray, DO, Pinellas Park, Florida
  - ACRC-Dermatology, West Palm Beach, Florida
  - Mark A Knautz, MD, Marietta, Georgia
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Grekin Skin Institute, Warren, Michigan
  - Jack C Scott, MD, Edina, Minnesota
  - Central Dermatology, St Louis, Missouri
  - Craig L Leonardi, MD, St Louis, Missouri
  - PMG Research of Raleigh, LLC, Cary, North Carolina
  - Box Arthritis & Rheumetology of the Carolinas, Charlotte, North Carolina
  - Michael Joseph Noss, MD, Cincinnati, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Dermatology and Skin Surgery Center, PC, Exton, Pennsylvania
  - James Henry Kopp, MD, Anderson, South Carolina
  - PMG Research of Bristol, LLC, Bristol, Tennessee
  - Arlington Research Center, Inc., Arlington, Texas
  - Center for Clinical Studies TMC/ Museum District Office, Houston, Texas
  - Center for Clinical Studies, Houston, Texas
  - Center for Clinical Studies, Webster, Texas
- Center for Dermatology and Venerology Diseases, EOOD, Sofia City, Sofia, Bulgaria
- Canada (10):
  - Kingsway Clinical Research, Etobicoke, Ontario
  - Dermatology Center, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - Research by ICLS, Oakville, Ontario
  - Skin Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - Research Toronto, Toronto, Ontario
  - Probity Medical Research, Inc., Waterloo, Ontario
  - Windsor Clinical Research, Windsor, Ontario
- Chile (3):
  - Clinica Dermacross SA, Santiago
  - Centro Intrnacional de Estudios Clinicos- CIEC, Santiago
  - Antonio Guglielmetti, MD, Viña del Mar
- Croatia (2):
  - Naftalan, Special Hospital for Medical Rehabilitation, Ivanić-Grad
  - Clinical Hospital Centre "Osijek", Osijek
- Estonia (3):
  - Tartu University Hospital, Dermatology Clinic, Raja, Tartu
  - Innomedica OÜ, Tallinn
  - North Estonian Medical Centre Foundation Skin and Sexual Diseases Center, Tallinn
- Georgia (5):
  - Aleksandre Aladshvili Clinic LLC, Tbilisi
  - Tbilisi State Medical University Alexandre Aladashvili University Clinic, Tbilisi
  - Scientific/Research National Center of Dermatology and Venereology, Tbilisi
  - Health Institute LLC, Tbilisi
  - Medical Center Clto Ltd, Tbilisi
- Israel (4):
  - Department of Dermatology- Ha'Emek Medical Center, Afula
  - Meir Medical Center Dermatologic Clinic, Kfar Saba
  - Rabin Medical Center Department of Dermatology, Petah Tikva
  - Department of Dermatology Phototherapy and Day Care Center, Ramat Gan
- Italy (3):
  - Department of Clinical and Molecular Sciences Dermatologic Clinic, Ancona
  - Department of Internal Medicine and Medical Specialties Unit of Dermatology, Reggio Emilia
  - Istituto di Clinica Dermosifilopatica Univeristà Cattolica del S.Cuore, Rome
- Latvia (3):
  - Janis Kisis, MD, Jūrmala
  - Riga 1st Hospital Skin and Sexually Transmitted Diseases Clinical Centre, Riga
  - Kristine Berzina, MD, PhD, Riga
- PMSI Institute of Cardiology, Chisinau, Moldova
- Poland (9):
  - Zdrowie Osteo-Medic s.c., Bialystok
  - ClinicMed Badurski i wspólnicy Spółka Jawna, Bialystok
  - Centrum Badań Kliniccznych, Gdansk
  - Grażyna Pulka Specjalistyczny Ośrodek, "ALL-MED", Krakow
  - CenterMed Kraków Śp. z o. o., Krakow
  - Synexus Polska Sp. z o. o. Oddzial w Poznaniu, Poznan
  - Niepubliczny Zaklad Opieki Zdrowtnej "NASZ LEKARZ", Torun
  - Synexus Polska Śp. z o.o., Warsaw
  - Wojewodzki Szpital Specjalistyczny we Wrocławiu, Oddział Dermatologiczny, Wroclaw
- Russia (7):
  - Altay State Medical University, Barnaul
  - Moscow Scientific and Practical Center of Dermatovenereology and Cosmetology of the Public Health Department of Moscow, Moscow
  - Moscow State University and Dentistry named after Evdokimov, Moscow
  - Imc "Sogaz", Saint Petersburg
  - Olga Mikerina, MD, Saint Petersburg
  - Alliance Biomedical Group, Saint Petersburg
  - Clinic of Skin and Venereal Diseases of the Saratov State Medical University, Saratov
- DOST - Dermatovenerologicke oddelenie sanatorneho typu, Svidník, Slovakia
- South Africa (7):
  - Panorama Medical Centre, Room 136, Panorama, Cape Town
  - Medicross Pretoria West 1st Floor, Pretoria West, Pretoria
  - Zubar Fazal Ahmed Vawda. MD, Durban
  - The Park, Room 201, 2nd Floor, Pinelands
  - Synopsis Research cc, Rondebosch
  - Synexus Heiderberg Clinical Research Centre, Somerset West
  - Clinical Projects Research SA (PTY) Ltd., Worcester
- Ukraine (11):
  - Medical Center Private Enterprise "Dzerkalo", Dnipro
  - Ivano-Frankivsk National Medical Univeristy, Dept. of Dermatology and Venereology based on Ivano-Frankivsk Regional Clinical Dermatology and Venereology Dispensary, Ivano-Frankivsk
  - Municipal Healthcare Institution "Kharkiv City Dermatovenereological Dispensary #2, Kharkiv
  - Khmel'nytskyy Regional Dermatovenereological Dispensary, Khmelnytskyi
  - National Medical University named after O.O.Bohomolets, Dept. of Dermatology and Venereology based on Oleksandrivska Clinical Hospital of Kyiv City, Dept. of Dermatology, Kyiv
  - National Medical University named after Danyla Galytskoho, Dept. of Family Medicine and Dermatology, Venereology based on Dept. of Dermatovenereology of the clinical Hospital of Ukrainian State Border Guard Services, Lviv
  - Odesa National Medical University, Department of Dermatic and Venereologic Diseases based on Odesa Regional Dermatovenereological Dispensary, Odesa
  - Municipal Institution "Rivne Regional Dermatology and Venereology Dispensary" of Rivne Regional Council, Rivne
  - Municipal Institution of Ternopil Regional Council Ternopil Regional Clinical Dermatovenereological Dispensary, Ternopil
  - Diagnostic and Treatment Dermatology and Gynecology Center, Uzhhorod
  - Municipal Institution "Zaporizhzhya Regional Dermatology and Venereology Clinical Dispensary" of Zaporizhzhya Regional Council, Zaporizhzhya

RESULTS

PARTICIPANT FLOW:
Groups:
- CHS-1420: CHS-1420 40mg 2 doses at Week 0/Day 0 then 1 dose every 2 weeks starting at Week 1 for 23 weeks. At Week 24 subjects will continue on to CHS-1420 open label until study end.
  CHS-1420
- Humira (Adalimumab) Reassigned to CHS-1420: Adalimumab (Humira) 40mg 2 doses at week 0/Day 0, then 1 dose every 2 weeks starting at Week 1 until Week 15. At Week 16 subjects initially randomized to adalimumab will be reassigned (1:1) to CHS-1420 40mg dose every 2 weeks for weeks 17-23. At week 24 subjects will switch to CHS-1420, 1 dose 40mg every 2 weeks, open label until study end.open label until study end.
  Adalimumab
  CHS-1420
- Humira (Adalimumab): Adalimumab (Humira) 40mg 2 doses at week 0/Day 0, then 1 dose every 2 weeks starting at Week 1 until Week 15. At Week 16 subjects initially randomized to adalimumab will be reassigned (1:1) to continue adalimumab treatment, 1 dose 40mg every 2 weeks for weeks 17-23. At week 24 subjects will switch to CHS-1420, 1 dose 40mg every 2 weeks, open label until study end..
  Adalimumab
  CHS-1420
Period: Overall Study
Arm/Group | CHS-1420 | Humira (Adalimumab) Reassigned to CHS-1420 | Humira (Adalimumab)
Started | 274 | 135 | 136
Completed | 220 | 101 | 117
Not Completed | 54 | 34 | 19

BASELINE CHARACTERISTICS:
Groups:
- Humira (Adalimumab) Reassigned to CHS-1420: Adalimumab (Humira) 40mg 2 doses at week 0/Day 0, then 1 dose every 2 weeks starting at Week 1 until Week 15. At Week 16 subjects initially randomized to adalimumab will be reassigned (1:1) to CHS-1420 40mg dose every 2 weeks for weeks 17-23. At week 24 subjects will switch to CHS-1420, 1 dose 40mg every 2 weeks, open label until study end.
  Adalimumab
  CHS-1420
- Humira (Adalimumab): Adalimumab (Humira) 40mg 2 doses at week 0/Day 0, then 1 dose every 2 weeks starting at Week 1 until Week 15. At Week 16 subjects initially randomized to adalimumab will be reassigned (1:1) to continue adalimumab treatment, 1 dose 40mg every 2 weeks for weeks 17-23. At week 24 subjects will switch to CHS-1420, 1 dose 40mg every 2 weeks, open label until study end.
  Adalimumab
  CHS-1420
- Total: Total of all reporting groups
Arm/Group | CHS-1420 | Humira (Adalimumab) Reassigned to CHS-1420 | Humira (Adalimumab) | Total
Number analyzed (Participants) | 274 | 135 | 136 | 545
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 256 | 124 | 127 | 507
  >=65 years | 18 | 11 | 9 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 31 | 38 | 151
  Male | 192 | 104 | 98 | 394

OUTCOME MEASURES:

1. Primary Outcome: Difference Between the Percentage of Subjects in Each Treatment Group Achieving a 75% Improvement in Psoriasis Area and Severity Index (PASI-75) at Week 12
Description: The efficacy success criterion was the equivalence between CHS-1420 and Humira at Week 12. Equivalence was based upon 2-sided 95% confidence interval (CI) for the difference between the proportions of subjects in the CHS-1420 and Humira groups achieving PASI-75 at Week 12. If the 95% CI lay entirely within the interval (-15%, 15%), equivalence was established.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Humira (Adalimumab): Adalimumab (Humira) 40mg 2 doses at week 0/Day 0, then 1 dose every 2 weeks starting at Week 1 until Week 15. At Week 16 subjects initially randomized to adalimumab will be reassigned (1:1) to CHS-1420 or continue adalimumab treatment, 1 dose every 2 weeks for weeks 17-23. At week 24 subjects will switch to CHS-1420 open label until study end.
  CHS-1420
  Adalimumab
Arm/Group | Humira (Adalimumab) | CHS-1420
Number analyzed (Participants) | 271 | 274
Participants | 203 | 211

ADVERSE EVENTS:
Groups:
- Treatment Period 1: CHS-1420: CHS-1420 40mg, 2 doses at Week 0/Day 0 then 40 mg, 1 dose every 2 weeks starting at Week 1 until Week 15
- Treatment Period 1: Humira (Adalimumab): Adalimumab (Humira) 40mg, 2 doses at Week 0/Day 0 then 40 mg, 1 dose every 2 weeks starting at Week 1 until Week 15.
- Treatment Period 2: CHS-1420/CHS-1420: At week 16 subjects initially randomized to CHS-1420 will continue CHS-1420 treatment 40 mg, 1 dose every 2 weeks starting at Week 16 to Week 24
- Treatment Period 2: Humira/CHS-1420: At Week 16 subjects initially randomized to Humira (adalimumab) will be reassigned to CHS-1420 treatment 40 mg, 1 dose every 2 weeks starting at Week 16 to Week 24
- Teatment Period 2: Humira/Humira: At Week 16 subjects initially randomized to Humira (adalimumab) will continue adalimumab treatment 40 mg, 1 dose every 2 weeks starting at Week 16 to Week 24
- Treatment Period 3: Open Label CHS-1420 Extension: At week 24 all subjects will switch to CHS-1420 treatment 40 mg, 1 dose every 2 weeks, open label, starting at week 24 until study end
Arm/Group | Treatment Period 1: CHS-1420 | Treatment Period 1: Humira (Adalimumab) | Treatment Period 2: CHS-1420/CHS-1420 | Treatment Period 2: Humira/CHS-1420 | Teatment Period 2: Humira/Humira | Treatment Period 3: Open Label CHS-1420 Extension
All-Cause Mortality (participants affected / at risk) | 0/274 | 0/271 | 0/255 | 0/126 | 0/130 | 1/474
Serious Adverse Events (participants affected / at risk) | 4/274 | 6/271 | 4/255 | 3/126 | 1/130 | 4/474
Other Adverse Events (participants affected / at risk) | 41/274 | 38/271 | 0/255 | 0/126 | 0/130 | 0/474
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period 1: CHS-1420 (N=274) | Treatment Period 1: Humira (Adalimumab) (N=271) | Treatment Period 2: CHS-1420/CHS-1420 (N=255) | Treatment Period 2: Humira/CHS-1420 (N=126) | Teatment Period 2: Humira/Humira (N=130) | Treatment Period 3: Open Label CHS-1420 Extension (N=474)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic and obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congenital Cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period 1: CHS-1420 (N=274) | Treatment Period 1: Humira (Adalimumab) (N=271) | Treatment Period 2: CHS-1420/CHS-1420 (N=255) | Treatment Period 2: Humira/CHS-1420 (N=126) | Teatment Period 2: Humira/Humira (N=130) | Treatment Period 3: Open Label CHS-1420 Extension (N=474)
Nasopharyngitis (Infections and infestations) | 24 (24) | 24 (24) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 17 (17) | 14 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT02489227/Prot_SAP_001.pdf